CLINICAL TRIAL: NCT03876561
Title: "Impact of Pelvic Floor Prehabilitation Using Biofeedback on the Severity of the Low Anterior Resection Syndrome in Patients Undergoing a Total Mesorectal Excision for Rectal Cancer"
Acronym: CONTICARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC16_0459
Record Dates: First submitted 2019-02-07; First posted 2019-03-15 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): The systematic pelvic floor prehabilitation will start 4 weeks before stoma closure and will include 1 sessions per week before stoma closure and 1 sessions per week during 6 weeks following stoma closure. Complementary sessions are allowed if necessary.
  Interventions: Procedure: Pelvic floor prehabilitation
- No intervention (No Intervention): No pelvic floor prehabilitation will be proposed before stoma closure. The pelvic floor prehabilitation will be proposed to patients suffering from LARS

INTERVENTIONS:
Procedure: Pelvic floor prehabilitation — The systematic pelvic floor prehabilitation will start 4 weeks before stoma closure and will include 1 session per week before stoma closure and 1 session per week during 6 weeks following stoma closure. The prehabilitation will be performed according to a predefined protocol based on a biofeedback strategy.
  Other Names: Preoperative rehabilitation
  Arms: Prehabilitation

SUMMARY:
There is currently no specific treatment and only few measures to prevent the low anterior resection syndrome (LARS). The LARS often results in a severe alteration of quality of life. This study is designed to assess pelvic floor prehabilitation using biofeedback in the prevention of LARS following total mesorectal excision for cancer. The pelvic floor rehabilitation with biofeedback has already been tested postoperatively in patients suffering from LARS with heterogeneous results. However, this rehabilitation has never been evaluated in the prevention of LARS.

The prehabilitation is an innovative concept currently evaluated in the prevention of functional complications following orthopedic surgery and also prostate surgery. In high-risk abdominal surgery, cardiopulmonary prehabilitation offers satisfying results in terms of morbidity and mortality rates. This study will be the first to assess pelvic floor prehabilitation in the prevention of LARS.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old
* Total mesorectal excision with colorectal or coloanal anastomosis protected by an ileostomy or a colostomy for rectal cancer
* Absence of anastomotic leakage or stenosis
* Informed consent to participate in the study
* Social security insurance affiliation

Exclusion Criteria:

* History of anal incontinence and/or fecal urgency and/or chronic diarrhea requiring a specific treatment before rectal cancer management
* Absence of ileostomy or colostomy
* Anastomotic leakage
* Sensorial or cognitive disorders impeding pelvic floor rehabilitation exercise
* Pregnant women
* Minors
* Adults under guardianship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Severity of Low Anterior Resection Syndrome Score (LARS score) | 6 months following stoma closure
  questionnaire assessing the five symptoms of the Low Anterior Resection Syndrome : fecal incontinence, gas incontinence, stool frequency, stool clustering and urgency.Total score is reported (minimum score :0 / maximal score : 42)

SECONDARY OUTCOMES:
Severity of fecal incontinence symptoms evaluated by the dedicated and validated score : Jorge and Wexner score | 6 months following stoma closure
  questionnaire to assess the severity of fecal incontinence symptoms, including stool frequency, stool and gas leakage, social impact and the frequency of pads.a total score is reported (minimum score :0 / maximal score : 20)
Impact on quality of life evaluated by the dedicated and validated questionnaire | 6 months following stoma closure
  questionnaire quality of life to assess the global quality of life in patients suffering from colorectal cancer Total score is reported
Morbidity of pelvic floor prehabilitation using biofeedback. | 6 months following stoma closure
  Biofeedback prehabilitation requires a small rectal manometry probe. This outcome will evaluate the morbidity of the rectal introduction of the probe following a colorectal anastomosis.
Medico-economic impact of pelvic floor prehabilitation including the fecal incontinence related costs | 6 months following stoma closure
  The fecal incontinence related costs will be quantified by the data obtained from the social security insurance and the patients' estimation. The differential benefit of the pelvic floor prehabilitation will be correlated to the quality of life estimated by the QALYS using the EQ-5D questionnaire.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU Angers, Angers
  - APHP-Hôpital Beaujon, Clichy
  - CHD Vendée, La Roche-sur-Yon
  - Clinic Jules Verne, Nantes
  - CHU de Poitiers, Poitiers
  - CHU de Tours, Tours

REFERENCES:
- [Derived] Alexandra P, Noemie P, Solene SB, Jean-Benoit H, Riche VP, Odile C, Michel G, Guy V, Hamy A, Mehdi O, Yannick T, Jeremie H L, Amar A, Emeric A, Jean-Michel B, Bridoux V, Dumont F, June F, Alexandra J, Meurette G, Duchalais E. Evaluation of pelvic floor rehabilitation in the prevention of low anterior resection syndrome: Study protocol of the CONTICARE trial. Colorectal Dis. 2025 Mar;27(3):e70045. doi: 10.1111/codi.70045. PMID 40055837